CLINICAL TRIAL: NCT05388357
Title: Fully Automated Quantitative Coronary Angiography Versus Optical Coherent Tomography Guidance for Coronary Stent Implantation (FLASH): Multicenter, Randomized Controlled Non-Interiority Trial
Brief Title: AI Quantitative Coronary Angiography Versus Optical Coherent Tomography Guidance for Coronary Stent Implantation
Acronym: FLASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Korea Medical Device Development Fund (Unknown); Medipixel,Inc (Unknown)
Responsible Party: Principal Investigator, Jung-min Ahn, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMCCV2022-02
Record Dates: First submitted 2022-05-10; First posted 2022-05-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Coronary Vessels; Procedure PCI
Keywords: OCT, AI ,PCI
MeSH Terms: conditions — Ornithine Carbamoyltransferase Deficiency Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI -guided PCI (Experimental): based on AI-QCA measurement, a drug eluting stent of an appropriate size is inserted and then high-pressure balloon dilatation is additionally actively performed in all patients.
  Interventions: Other: Intervention Procedure: PCI
- OCT-guided PCI (Active Comparator): In the OCT group, the size of the stent is determined using intravascular optical coherence tomography, and balloon dilatation is additionally performed if necessary.
  Interventions: Other: Intervention Procedure: PCI

INTERVENTIONS:
Other: Intervention Procedure: PCI — Percutaneous Coronary Intervention

SUMMARY:
This study is to establish the primary hypothesis thatAI -QCA guided PCI is non-inferior to Optical coherence tomography-guided Percutaneous coronary intervention regarding minimal Stent area by Final OCT and Procedural MACE

DETAILED DESCRIPTION:
1. AI-QCA-assisted DES implantation

   After coronary angiography, AI-QCA software will be used to determine the lesion length and the reference vessel diameter in real time to determine the appropriate stent size for implantation. The procedure is performed as follows:
   1. Select the optimal projection angle providing the best view of the lesion.
   2. Provide sufficient nitroglycerin for vasodilation. If the lesion is severely stenotic, perform balloon angioplasty, followed by nitroglycerin supply.
   3. Perform AI-QCA to measure the length of the lesion and the inside diameter of the proximal and distal reference vessels.
   4. Determine the stent length and size according to the AI-QCA measurements. Select a stent that is 20% larger than the distal reference vessel diameter and that can provide coverage for both the proximal and distal reference vessels.
   5. Perform high-pressure balloon dilation after stent implantation, with the final balloon size being 20% larger than the distal and proximal reference vessel diameters.
   6. Perform a final coronary angiogram if no procedural complications are observed on the angiogram and stent expansion is confirmed.
   7. Perform a final OCT to measure the stent area (mm2), the primary efficacy endpoint.
   8. If significant suboptimal stent results, such as severe underexpansion, extensive strut malapposition, or major stent edge dissection, occur, additional procedures to correct them are permitted to ensure patient safety, although they are generally discouraged. (The primary endpoint will be assessed by OCT run before such correction.)
2. OCT guided DES implantation

After coronary angiography, OCT is performed to determine the appropriate stent size for implantation. After the stent procedure, OCT is performed again to check for an area that is smaller than the area of distal reference vessel and for sufficient dilatation. If necessary, high-pressure balloon dilation is performed to minimize residual stenosis. The procedure is performed as follows:

1. Select the optimal projection angle providing the best view of the lesion.
2. Provide sufficient nitroglycerin for vasodilation. If the lesion is severely stenotic, perform balloon angioplasty, followed by nitroglycerin supply.
3. Perform OCT to obtain pre-procedural images of the vessel. If there is a stenosis and OCT images cannot be obtained, perform OCT after adequate balloon angioplasty.
4. Determine the length and size of the stent to be implanted according to the OCT images. Select the stent size in consideration of the mean lumen diameter and mean external elastic lamina (EEL) diameter of the distal reference vessel. If the EEL is not observed, use a stent that is 0.25 mm larger than the mean lumen diameter. Select the length by measuring the length of the proximal and distal reference vessel segments on the OCT.
5. Perform high-pressure balloon dilation after stent implantation. Select the final balloon size by considering the inside diameters of the distal and proximal reference vessels and EEL diameter.
6. Perform OCT. If no procedure-related complications are observed and there is no underexpansion or malapposition of the stent, perform a final coronary angiogram. If procedure-related complications or underexpansion or malapposition of the stent is observed, correct it, and then perform a final OCT to measure the stent area (mm2), the primary efficacy endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Men or women at least 19 years of age
* Patients with typical symptoms or objective evidence of myocardial ischemia and eligible for coronary angioplasty.
* Subject with severe coronary artery disease undergoing PCI
* Written informed consent

Exclusion Criteria:

* Angiographic exclusion criteria 1) Left main lesion 2) Chronic total occlusion 3)Graft vascular lesion 4) Requiring two-stent techniques for coronary bifurcation lesions 5)Any lesion characteristics resulting in the expected inability to deliver OCT catheter to the lesion ( eg,tortuosity, moderate or severe vessel calcification)
* Acute or chronic renal dysfunction (Plasma creatinine 2.0mg/dL or more) except patients undergoing dialysis
* Primary coronary angioplasty in ST-elevation myocardial infarction(within 12-24 hours of symptom onset)
* Previous PCI with BVS
* LV dysfunction (LVEF) < 30%
* Hypersensitivity to DES and its components or there is a reason for prohibition (everolimus, cobalt, chromium, nickel, platinum, tungsten, acrylic and fluoro polymers)
* Patients who require surgery requiring discontinuation of antiplatelet drugs within 1 year of the procedure
* Life expectancy < 1 year for any disease
* Pregnancy or breast-feeding
* Patients unsuitable for enrollment judged by the Investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
Minimal Stent Area evaluated by OCT | 1hour
  Minimal Stent Area evaluated by OCT after stenting of the target lesion
Procedural complications | 24hours
  Procedural complications including angiographic dissection, perforation, or acute closure requiring active intervention after stent implantation

SECONDARY OUTCOMES:
Procedural success | 24hours
  Stent expansion (≥ 90%) in final OCT assessment and successful stent delivery without target-lesion failure in 24 hours
OCT endpoint | 24hours
  Stent expansion, stent malapposition, intra-stent tissue (plaque or thrombus) protrusion, untreated reference segment disease
Angiographic endpoint | 24hours
  Minimal lumen diameter at the stented segment, diameter stenosis at the stented segment, acute gain at the stented segment
Death | 6month
  All-cause death , Cardiac and non-Cardiac death
MI | 6month
  Any MI( periprocedural/spontaneous MI), Target vessel-MI and non-target vessel-MI
Stent thrombosis | 6month
  definite/probable
Revascularization | 6month
  Any revascularization,Target vessel and target lesion revascularization
Composite of event | 6month
  Composite of all-cause death, myocardial infarction, stent thrombosis, or revascularization
Quality of life score assessed by the EQ-5D | 6month
  The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
  EQ-5D: the minimum and maximum values are 5 and 25 respectively. EQ VAS: the minimum and maximum values are 0 and 100 respectively.
Quality of life score assessed by Health-related Quality of Life Instrument with 8 Items (HINT-8) | 6month
  HINT-8 was developed based on 4 health dimensions: physical, mental, social, and positive health dimensions. It consists of climbing stairs, endurance to pain, vitality, working, depression, memory, sleep, and happiness.
Cost-effective analysis | 6month
  Cost-effective analysis based on average treatment costs for two treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jung- min Ahn, Principal Investigator — Asan Medical Center
Locations (13):
- South Korea (13):
  - Sejong General Hospital, Bucheon-si
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu
  - GangNeung Asan Hospital, Gangneung
  - Seoul National University Bundang hospital, Gyeonggi-do
  - Soon Chun Hyang University Hospital Bucheon, Gyeonggi-do
  - Yougin Severance Hospital, Gyeonggi-do
  - Chungbuk National University Hospital, Jungbuk
  - Pusan National University Hospital, Pusan
  - Asan Medical Center, Seoul
  - Hanyang University Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim Y, Yoon HJ, Suh J, Kang SH, Lim YH, Jang DH, Park JH, Shin ES, Bae JW, Lee JH, Oh JH, Kang DY, Kweon J, Jo MW, Yun SC, Park DW, Kim YH, Park SJ, Park H, Ahn JM; FLASH Trial Investigators. Artificial Intelligence-Based Fully Automated Quantitative Coronary Angiography vs Optical Coherence Tomography-Guided PCI: The FLASH Trial. JACC Cardiovasc Interv. 2025 Jan 27;18(2):187-197. doi: 10.1016/j.jcin.2024.10.025. Epub 2024 Oct 30. PMID 39614852
- [Derived] Kim Y, Park H, Yoon HJ, Suh J, Kang SH, Lim YH, Jang DH, Park JH, Shin ES, Bae JW, Lee JH, Oh JH, Kang DY, Kweon J, Jo MW, Park DW, Kim YH, Ahn JM; FLASH Trial Investigators. Fully automated quantitative coronary angiography versus optical coherence tomography guidance for coronary stent implantation (FLASH): Study protocol for a randomized controlled noninferiority trial. Am Heart J. 2024 Sep;275:86-95. doi: 10.1016/j.ahj.2024.05.004. Epub 2024 May 7. PMID 38723880